CLINICAL TRIAL: NCT04673760
Title: Palliative Needs Assessment and Palliative Care in Primary Care: The PROAKTIV Study
Brief Title: The PROAKTIV Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); University of Bern (Other)
Responsible Party: Principal Investigator, Steffen Eychmüller, Prof. dr. med., Insel Gruppe AG, University Hospital Bern
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DFL Nr. 4887; SNCTP000003820 (Registry Identifier: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2020-11-03; First posted 2020-12-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Palliative Care
Keywords: palliative care; end of life care; home care services; primary care; primary care nursing; outpatient care; quality of healthcare; quality of life; advance care planning

STUDY DESIGN:
Intervention Model Description: Patients with a new medical indication for specialized palliative home care are assigned to intervention arm.
  Patients without a new indication for specialized palliative home care are controls .
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Structured specialized palliative home care (Experimental): Eligible specialist palliative home care teams provide ambulant specialised palliative care as usual
  Interventions: Behavioral: Specialized palliative home care
- Arm 2: No care of specialist palliative home care teams at study inclusion (No Intervention): No care from specialist palliative home care teams at study inclusion

INTERVENTIONS:
Behavioral: Specialized palliative home care — Specialist palliative home care teams will initiate care as usual, including managing a systematic and collaborative process of advance care planning with patients, family caregivers, GPs and SPITEX nurses using the "Betreuungsplan", information packages and regular case meetings. The GP was additionally provided with educational palliative care information by the study team.
  Arms: Arm 1: Structured specialized palliative home care

SUMMARY:
The overall objective of this study is to identify whether the systematic anticipation of highly structured specialized palliative home care into primary care influences the quality of care and care utilization. Quality of care focusses on the sense of security of patients and family caregivers, satisfaction with care of patients, family caregivers, general practitioners, home care nurses and specialized palliative care nurses, and availability and access to advanced directives. Health care utilization focus on the number of hospitalizations and the length of hospital stays.

DETAILED DESCRIPTION:
The University Center for Palliative Care from the Inselspital Bern conducts this monocentric mixed-methods controlled study and is responsible for informed consent.

Data consists of questionnaires of patients, their family caregivers, general practitioners, home care nurses and if involved specialized palliative home care nurses. Patients and their family caregivers will fill out baseline questionnaires and follow-up questionnaires at 2, 8, 16 and 24 weeks. Patient follow-up will end if the patient dies or the study ends. Family caregivers will be asked to fill out a questionnaire two months after the patient's death.

General practitioners, home care nurses and specialised palliative home care nurses will fill out questionnaires after the patient's death or at the end of the study. Patient survival data will be collected from administrative health data after the end of the study.

Additionally, a nested qualitative study with semi-structured qualitative interviews with patients, family caregivers and care providers will provide an in-depth understanding of preferences, needs, experiences from this phase of life.

ELIGIBILITY:
Patients inclusion criteria:

* 18 years or older
* Able to read and understand German
* Able to fill out questionnaires with only minimal assistance
* Live in the catchment area of SPHC
* Positive screening on the palliative care screening tools
* Expected survival time of approximately six months or less
* Have a GP (or GP medical substitute)
* Registered with Spitex care
* Wish to live at home as long as possible (no plans for long term nursing home uptake)
* Written informed consent

Patients exclusion criteria:

* Planned discharged from hospitals to institutions (e.g. other hospitals, rehabilitations, nursing homes)
* Live permanently in nursing homes
* Cognitive impairments that make it impossible to follow the study (e.g. psychological disorders, dementia, loss of judgement).

Family caregivers inclusion criteria:

* 18 years or older
* Able to read and understand German
* Familiar with the care situation patient
* Written informed consent

Specialized palliative home care team:

* Provide care in German speaking part of canton Bern
* 24/7-availability of specialized palliative care
* Specialized palliative care team including nurses and consulting physician with specialized palliative care certification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Sense of security of patients | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire Sense of Security in Care - Patients' Evaluation (SEC-P), This questionnaire has 3 subscales namely, the Care Interaction scale; the Identity scale and the Mastery scale. Higher score indicate a higher level of sens of security at home of the patient.

SECONDARY OUTCOMES:
Number of patients who define advance directives | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire
Access to advance directives of the patients for the ambulant care providers | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire
Satisfaction with care of patient | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire Modified FAMCARE Scale P16. 16 Questions on care with answers (Likert-type scale 1 to 5) ranging from "very satisfied with care" to "very dissatisfied with care"
Satisfaction with care of GP | From date of baseline measurement of patient to study completion, an average of 6 months, or shorter if patient deceases
  Measured by questionnaire

OTHER OUTCOMES:
Health care utilization | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire
Health care costs | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by administrative health care data
Sense of security of family caregivers | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire
Satisfaction with care of family caregivers | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire FAMCARE-2 Scale. 17 questions on care with answers ( Likert-type scale 1 to 5) ranging from "very satisfied with care" to "very dissatisfied with care".
Satisfaction with care of home care nurses | From the date of baseline measurement of patient to study completion, an average of 6 months, or shorter if patient deceases
  Measured by questionnaire
Performance Status of patient | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire , ECOG Scale of performance status.Grading 1 to 4 and higher score indicates lower performance status.
Quality of life of patient | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire Functional Assessment of Chronic Illness Therapy - Palliative Care 14 Item Version (FACIT-Pal-14). (5 point Likert-type scale)
Therapeutic alliance between patients and their home care team | From 2 months before the date of baseline measurement (retrospectively), to six months after the baseline measurement (prospectively).
  Measured by questionnaire The Human Connection Scale (THC) measures the extent to which patients felt a sense of mutual understanding, caring, and trust with their GP, (specialized palliative) home care nurses ( Likert-type scale 1 to 5)

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Eychmüller, Prof. dr., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No